CLINICAL TRIAL: NCT01685827
Title: Efficacy and Safety of Fexinidazole Compared to Nifurtimox-Eflornithine Combination Therapy (NECT) in Patients With Late-stage Human African Trypanosomiasis (HAT) Due to T.b. Gambiense: Pivotal, Non-inferiority, Multicentre, Randomised, Open-label Study
Brief Title: Pivotal Study of Fexinidazole for Human African Trypanosomiasis in Stage 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DNDiFEX004
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Human African Trypanosomiasis (HAT); Sleeping Sickness
MeSH Terms: conditions — Trypanosomiasis, African | interventions — fexinidazole; Nifurtimox; Eflornithine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NECT (Nifurtimox Eflornithine Combination Therapy) (Active Comparator): * Nifurtimox tablets will be given orally three times a day, at the daily dose of 15 mg/kg/day, for 10 days.
  * Eflornithine (400 mg/kg/day) will be given twice daily for 7 days, as a 2-hour IV infusion.
  Interventions: Drug: Nifurtimox; Drug: Eflornithine
- Fexinidazole (Experimental): Fexinidazole, 600 mg tablets given by oral route, after the main daily meal (within 30 minutes from the start of the meal), at the daily dose of:
  * 1 800 mg (3 tablets) once a day for 4 days,
  * Followed by 1 200 mg (2 tablets) once a day for 6 days. Total duration of treatment will be 10 days.
  Interventions: Drug: Fexinidazole

INTERVENTIONS:
Drug: Fexinidazole
  Arms: Fexinidazole
Drug: Nifurtimox
  Other Names: Lampit
  Arms: NECT (Nifurtimox Eflornithine Combination Therapy)
Drug: Eflornithine
  Other Names: Ornidyl
  Arms: NECT (Nifurtimox Eflornithine Combination Therapy)

SUMMARY:
This clinical trial is designed to prove the efficacy and safety of Fexinidazole as an oral treatment for human african trypanosomiasis in advanced stage. The Fexinidazole is compared to reference treatment NECT. The trial will try to demonstrate that Fexinidazole is not inferior to NECT treatment.

DETAILED DESCRIPTION:
Human African Trypanosomiasis (HAT) is a life-threatening and neglected disease.

Few treatment options are currently available for stage 2 (meningo-encephalitic stage) HAT, with NECT being the most commonly used one since 2010. Though NECT represents a significant improvement over current therapies, it is still far from ideal given the environment in which HAT patients live (remote, poor areas with little health infrastructure, if any, and difficult logistics). There is an urgent need for less toxic and more easily manageable compounds to treat this fatal disease.

Fexinidazole is a 2-5-nitroimidazole, formulated for oral administration, which has been shown to possess in vitro and in vivo activity against both T. b. rhodesiense and T. b. gambiense parasites.

Predicted CSF concentrations reached target levels after repeated dosing. Its efficacy and safety must now be tested in patients with stage 2 HAT.

ELIGIBILITY:
Inclusion Criteria:

* 15 years old or more
* Male or female
* Able to ingest at least one complete meal per day (or at least one Plumpy'Nut® sachet)
* Karnofsky index>50 (see Appendix 2 - Karnofsky Scale; p81)
* Parasitologically confirmed late-stage African trypanosomiasis infection with T. b. gambiense in the blood and/or lymph and/or CSF, attested by mobile team report (with detail of exams performed and values of WBC measured in CSF) or done at the study centre. If parasitologically negative in CSF, WBC >20/µl detected in the CSF to document stage 2 infection.
* Having a permanent address and able to comply with follow-up visit schedule
* Signed Informed Consent Form

Exclusion Criteria:

* Severely malnourished patients, defined as having a BMI < 16.
* Patients unable to take oral medication.*
* Pregnancy or lactation
* Active clinically relevant medical conditions that, in the Investigator's opinion, may jeopardize subject safety or interfere with participation in the study, including but not limited to significant liver or cardiovascular disease, active documented or suspected infection, CNS trauma or seizure disorders, coma or altered consciousness.
* Severely deteriorated general condition, such as cardiovascular shock, respiratory distress, or terminal illness.
* Any condition which compromises ability to communicate with the Investigator as required for the completion of this study.
* Any contraindication to imidazole products (known hypersensitivity to imidazoles) and NECT (known hypersensitivity to eflornithine).
* Patients previously treated for HAT.
* Patients previously enrolled in the study.
* Follow-up expectable difficulties (migrants, refugees, traders, etc.).
* History of alcohol abuse or any drug addiction.
* Clinically significant abnormal laboratory value
* Pregnancy
* Unstable ECG abnormalities
* QTcF≥ 450 msec in resting position (confirmed by 2 measurement).
* Patients not tested for malaria and/or treated adequately for this infection
* Patients not treated adequately for soil transmitted helminthic diseases

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2012-10; Primary Completion 2016-11-11 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
success or failure at 18 months FU visit | 18 months after treatment
  The primary endpoint is the outcome (success or failure) at the test of cure (ToC) visit 18 months after the end of treatment (EOT) adapted from WHO criteria.
  Success at 18 months is:
  * Either cure:
    * patient alive,
    * AND with no evidence of trypanosomes in any body fluid,
    * AND 20 or less WBC/µl CSF
  * Or Probable cure:
    * Patient with no parasitological evidence of relapse in blood and lymph
    * AND who refuses lumbar puncture OR whose CSF sample is haemorrhagic without trypanosomes
    * AND whose clinical condition is satisfactory (without clinical symptom or signs) OR whose clinical status is unlikely to be due to HAT

SECONDARY OUTCOMES:
Safety endpoint | 18 days - observation period
  Occurrence of any grade (all grades combined) adverse events during the observation period (D1-18) including:
  * any worsening of clinical symptoms listed in the inclusion checklist of symptoms and signs,
  * laboratory abnormalities of grade ≥ 2
  * Occurrence of grade ≥ 3 adverse events during the observation period
  * Occurrence of drug-related adverse events (grade ≥ 3 and any grade) during the observation period
Safety endpoint | 24 months
  Occurrence of any serious adverse events from first drug intake to the end of follow-up period (18 months), and from M18 to M24.
Pharmacokinetics endpoint | from D8 to D12 after first dosing
  Whole blood and CSF concentrations of fexinidazole, M1, M2 and PK parameters derived from a model of population PK data.
QT evaluation | D0 - D4 - D10
  recording of triplicates ECG

CONTACTS AND LOCATIONS:
Overall Officials: Victor KANDE, MD, Principal Investigator — HAT National Control Program in DRC
Locations (10):
- Batangafo, Batangafo, Central African Republic
- Bagata Hospital, Bagata, Bandundu, Democratic Republic of the Congo
- Republic of the Congo (8):
  - Masi Manimba Hospital, Masi Manimba, Bandundu - DRC
  - Vanga Hospital, Vanga, Bandundu - DRC
  - HGR (General Reference Hospital) Bandundu, Bandundu, Bandundu
  - HGR Mushie hospital, Mushie, Bandundu
  - CRT (Centre de Réference et de Traitement) Dipumba, Dipumba general hospital, Mbuji Mayi, East Kasai
  - HS Katanda hospital, Katanda, Kasaï Oriental
  - HGR ISANGI hospital, Isangi, Province Orientale
  - Dingila, Dingila

REFERENCES:
- [Derived] Mesu VKBK, Kalonji WM, Bardonneau C, Mordt OV, Blesson S, Simon F, Delhomme S, Bernhard S, Kuziena W, Lubaki JF, Vuvu SL, Ngima PN, Mbembo HM, Ilunga M, Bonama AK, Heradi JA, Solomo JLL, Mandula G, Badibabi LK, Dama FR, Lukula PK, Tete DN, Lumbala C, Scherrer B, Strub-Wourgaft N, Tarral A. Oral fexinidazole for late-stage African Trypanosoma brucei gambiense trypanosomiasis: a pivotal multicentre, randomised, non-inferiority trial. Lancet. 2018 Jan 13;391(10116):144-154. doi: 10.1016/S0140-6736(17)32758-7. Epub 2017 Nov 4. PMID 29113731
- See also: Sponsor Website — http://www.dndi.org